CLINICAL TRIAL: NCT02900066
Title: Filter Paper Blood Spots Collected During Fever as a Source for Post-travel Diagnosis of Arboviral and Rickettsial Infections in a Cohort of Travelers
Brief Title: Filter Paper Blood Spots Collected During Fever as a Source for Post-travel Diagnosis in Travelers
Acronym: JOKA-II
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: B-300201627244
Record Dates: First submitted 2016-03-16; First posted 2016-09-14 (Estimated); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Fever
Keywords: fever; traveler; arbovirus; rickettsia; malaria; filter paper; diagnosis
MeSH Terms: conditions — Fever; Malaria; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — sera, capillary blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is part of a larger prospective cohort study (JOKA), designed to study febrile illness occurring during a travel to the tropics, as well as the evaluation of the clinical use of malaria rapid diagnostic tests (RDT) by travelers or their peers during travel, as a decision aid for the management of febrile illness in the tropics.

Filter paper blood spots and paired serology are used in addition to routine post-travel evaluation, to study the incidence and etiological spectrum of febrile illness occurring during travel to the tropics.

The study will yield valuable and prospective data of incidence rate, the clinical and etiological spectrum, clinical course and outcome of febrile illness during (and post-)travel in a prospective cohorts of travelers. This knowledge may lead to better pre-travel advice.

DETAILED DESCRIPTION:
Objectives:

To study the incidence etiological spectrum of febrile illness occurring during a travel to the tropics, as well as clinical course, care, treatment and outcome of these febrile illness episodes.

Design: Prospective cohort study of febrile illness in international travelers Population: Travelers who are going to destinations in the tropics (South-East Asia (SEA), Sub-Saharan Africa (SSA) and South America (SCA)) for 3 weeks or longer will be invited to participate and, after obtaining informed consent, recruited in the study protocol(s) at the time of planning departure (directly at the ITM or through travel/ humanitarian relief organizations).

Methods:

Participants will be offered pre-, per- and post-travel consultation as explained below (Inclusion through ITM)

1. Pre-travel consultation at a certified travel clinic will systematically be recommended; this consultation will include:

1. routine travel advice directed at travel destination, (including vaccinations and prescription for anti-malarial chemoprophylaxis according to current recommendations, details of which are published at www.reisgeneeskunde.be and
2. the following research-related activities.

   * Briefing sessions on the topic "Fever in The Tropics" by an ITM physician (during this session the differences between fever at home and in the tropics will be addressed and the importance of consulting a local doctor will be stressed).
   * Collection and recording of demographic, clinical and travel data.
   * Sampling of a baseline serum sample (for paired pre- and post-travel diagnostic analysis).
   * Training of travelers, peers and travel guides to blot capillary blood on a filter paper (training is a prerequisite for study participation).
   * Provision of study materials (study diary/apps, malaria kits, thermometer, …) and written instructions for use during travel if fever occurs (see below)

     2. During travel
   * In case of any illness (associated with fever or not), the traveler will record symptoms in the study diary.
   * If fever is documented (axillary temperature ≥ 37.8°C - or in case a thermometer is not immediately available, fever sensation in association with sweats or chills)- blood from a finger prick will be collected for blotting onto filter paper (BFP) by trained travelers or peers.
   * All febrile travelers are advised to seek medical attendance as they would do when not participating in the study.
   * The final decision to use standby emergency treatment malaria treatment (SBET) is made by the study participant, in accordance with precise and written instructions.
   * The study team (Tropical medicine experts at ITM) will be available for teleconsultation by Email or Telephone, and will provide medical advice within 12 hours. Note: contacting the ITM study team is an option, but should not cause delay in treating suspected malaria.
   * Study participants will collect all relevant data related to the (outcome of the) illness episode (duration of symptoms, consultation of a health practitioner, admission/duration of stay in a hospital, treatment received and timing, repatriation)

     3. Post-travel consultation will be scheduled for all study participants who experience(d) any illness (febrile or not) within a week after travel- sooner if the medical condition requires so- and for those who have no complaints but do seek post-travel health evaluation.
   * A structured clinical evaluation will be performed by an expert in travel medicine and will be recorded in the database. Laboratory evaluation will include hematological, biochemical and microbiological/parasitological analysis
   * Used BFPs (i.e. in case of febrile illness during travel) will be collected for confirmation of the test result by Polymerase Chain Reaction (PCR). A diagnostic protocol/ algorithm will be developed for use the BFPs as a source for post-travel diagnosis of arboviral/ rickettsial infection by PCR.

     * Data analysis : All data (demographic, geographic, clinical, laboratory and final diagnosis) will be recorded in an encoded database. Descriptive and inferential statistics as appropriate, STATA 14.
     * Sample size: n= 350 fever cases; at an incidence of fever of 8% a cohort of 4400 (healthy) travelers will be recruited over 30 months (Feb 2016 - Aug 2018).
     * Endpoints:
   * Incidence rates for malaria and arboviral/ rickettsial infections (by paired serology and post-travel PCR on BFP) per travel destination.
   * Clinical course and outcomes of (self-)management of febrile illness during travel. (Clinical spectrum of disease, incidence rates of febrile illnesses; duration of fever and other symptoms, management (self-treatment, consultation, admission), type of treatment (symptomatic/empiric/targeted if RDT malaria positive), final outcome (change of travel plans, repatriation, hospitalization as a result of illness during travel).

Expected results and relevance: The study will yield valuable and prospective data of incidence rate, the clinical and etiological spectrum, clinical course and outcome of febrile illness during (and post-)travel in a prospective cohorts of travelers. This knowledge may lead to better pre-travel advice.

ELIGIBILITY:
Inclusion Criteria:

* Residing in Belgium.
* Attend a briefing session on the topic "Fever in The Tropics" by an ITM physician.
* Able to comply with study procedures:

  * Carry and complete a study diary in case of illness
  * Be trained to collect BFP OR
  * Travel with anyone who has been trained
* Willing and able to provide written informed consent.
* Adults fulfilling all criteria and volunteer to have their BFP collected by their trained peers during travel, may be included for analysis after obtaining informed consent upon post-travel evaluation.

Exclusion criteria:

* Unable to comply with study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons intending to travel to Asia, Africa, or America for a minimum duration of 3 weeks
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of etiological diagnoses in febrile travelers as assessed by post hoc clinical evaluation | up to 6 months of follow-up per individual traveler
  PCR analysis will be directed by antibody detection in paired sera, and post-travel clinical evaluation

SECONDARY OUTCOMES:
Clinical outcome of febrile illness during travel | up to 6 months of follow-up per individual traveler
  Final clinical outcome per diagnosis (change of travel plans, repatriation, hospitalization as a result of illness during travel, death).
incidence of etiological diagnoses of fever expressed as risk per person- year of travel per region traveled | up to 6 months of follow-up per individual traveler
Time from start of travel to development of fever by self-reporting | up to 6 months of follow-up per individual traveler
duration of symptoms by self-reporting in a structured study diary | up to 6 months of follow-up per individual traveler
Type of treatment per diagnosis reported in a structured study diary | up to 6 months of follow-up per individual traveler
  symptomatic/ empiric/ targeted upon diagnosis abroad

CONTACTS AND LOCATIONS:
Overall Officials: Jan Jacobs, MD PhD, Study Chair — Institute of Tropical Medicine, Antwerp, Belgium
Locations (1):
- ITM, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huits R, Van Den Bossche D, Eggermont K, Lotgering E, Feyens AM, Potters I, Jacobs J, Van Esbroeck M, Cnops L, Bottieau E. Incidence of Zika virus infection in a prospective cohort of Belgian travellers to the Americas in 2016. Int J Infect Dis. 2019 Jan;78:39-43. doi: 10.1016/j.ijid.2018.10.010. Epub 2018 Oct 24. PMID 30368020
- Available data/document: Individual Participant Data Set — https://doi.org/10.1016/j.ijid.2018.10.010 — The data supporting the findings of this study/publication are retained at the Institute of Tropical Medicine, Antwerp and will not be made openly accessible due to ethical and privacy concerns. Data can however be made available after approval of a motivated and written request to the Institute of Tropical Medicine at ITMresearchdataaccess@itg.be/.